CLINICAL TRIAL: NCT01227343
Title: Sex, GABA and Nicotine: A 1H-MRS Study
Brief Title: Nicotine and Brain Imaging Research Study
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 810278
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Nicotine
Keywords: Gender differences; nicotine; cigarette smoking habits; behavior changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, plasma, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Female Smokers: Healthy females who smoke 10-30 cigarettes per day for the past 2 years and meet criteria for nicotine dependence.
- Female Non-smokers: Healthy females who do not currently smoke cigarettes.
- Male Smokers: Healthy males who smoke 10-30 cigarettes per day for the past 2 years and who meet criteria for nicotine dependence.
- Male - Non-Smokers CLOSED: WE ARE NO LONGER RECRUITING MALE NON-SMOKERS

SUMMARY:
The aim of this study is to assess the impact of smoking on cortical GABA levels in males and females. Using magnetic resonance spectroscopy (MRS), we will examine the impact of sex and menstrual cycle phase on brain neurochemistry in healthy smokers and non-smokers. We hypothesize that female, but not male, smokers will have reduced cortical GABA levels compared to their non-smoking, sex-matched counterparts.

DETAILED DESCRIPTION:
The purpose of this study is to measure and compare gamma-aminobutyric acid (GABA) levels in the occipital cortex of a group of healthy smoking and non-smoking women and men ages 18-50. We will recruit women with regular menstrual cycles so that we can assess premenstrual impact of smoking cessation in that population and compare GABA level concentrations across all groups. Although there are several note-worthy differences between male and females in regard to smoking behavior, ultimately none are as worrisome as the disparity in ability to quit smoking. While multiple explanations for why women are less successful in their abstinence attempts have been proffered, the observation that women are more likely to experience emergence of depressive symptoms during smoking cessation, a known risk factor for relapse, may be the most important contributor to this sex-specific recidivism. Several lines of evidence suggest that nicotine modulation of GABA may play an important role in this interplay between sex, depression, and smoking recidivism.

ELIGIBILITY:
Inclusion Criteria:

Women ages 18-50 will be eligible for this study if they:

* Meet DSM-IV criteria for nicotine dependence for at least the past 2 years;
* Smoke 10-30 cigarettes per day for the past two years;
* Have clear urine toxicology screen upon recruitment and a plasma cotinine level of > 210 ng/ml;
* Have an expired CO (carbon monoxide) level of > 11ppm;
* Have regular menstrual cycles 24 to 36 days in length;
* Do not have an elevated follicular stimulating hormone (FSH) >20 (>20 is potentially indicative of menopause and would be an exclusion criterion);
* Have no history of major depressive disorder, generalized anxiety disorder, and or panic disorder within the last three years according to the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-NP) (First et al., 1995); a history of major depressive disorder, generalized anxiety disorder, and or panic disorder greater than 3 years ago, but now resolved according to the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-NP) (First et al., 1995), is allowed;
* Have no substance abuse disorders (this includes alcohol, prescription, and illicit substances) within the last three years other than nicotine dependence according to the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-NP) (First et al., 1995);
* Subject has history of substance abuse disorders (this includes alcohol, prescription, and illicit substances) >3 years ago but the period of abuse did not last more than 5 years according to the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-NP) (First et al., 1995);
* No history of clinically interfering premenstrual mood changes;
* Are able to give written informed consent;
* Are fluent in written and spoken English.

Exclusion Criteria:

* A psychiatric history of psychotic disorders, bipolar disorder, obsessive compulsive disorder, eating disorders, post-traumatic stress disorder, phobias (includes simple and specific phobias) and Axis II disorders;
* A history of serious medical or neurological illness, including (but not limited to) major cardiovascular disease, severe hypertension, intracranial mass lesions, seizure disorder, severe hepatic or renal disease, unstable endocrine or metabolic disease, and unstable hematologic disease;
* Use of psychotropic medication within the previous 12 months;
* Hazardous drinking in the previous 90 days defined as more than 7 drinks per week for women and more than 14 drinks per week for men, or more than 3 and 4 drinks in a single day for women and men, respectively;
* Hamilton Rating Scale for Depression (HAM-D; Hamilton, 1960) score >12;
* Mini-Mental State Examination (MMSE) >24;
* Use of steroidal contraceptives or hormone treatment within the previous 4 months;
* Current pregnancy;
* History of claustrophobic symptoms;
* Metallic implants.

For Healthy Non-Smoking Females:

Same inclusion/exclusion criteria for smoking females with the exception of the criteria related to smoking.

For Smoking Males:

Same inclusion/exclusion criteria for smoking females with the exception of the criteria related to menstrual cycle, conception, and FSH.

For Healthy Non-Smoking Males:

Same inclusion/exclusion criteria for smoking males with the exception of the criteria related to smoking.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women and men from the greater Philadelphia and surrounding areas who are ages 18-50 will be considered for enrollment into this study.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
To estimate and compare the impact of smoking on cortical GABA levels in male and female smokers and non-smokers. | 3-10 weeks
  Preliminary findings suggest that nicotine's effects on cortical GABA levels vary by sex with women experiencing the greatest smoking-induced alterations in cortical GABA levels. We hypothesize that female, but not male, smokers will have reduced cortical GABA levels compared to their non-smoking, sex-matched counterparts.

SECONDARY OUTCOMES:
To measure occipital cortex GABA concentrations in healthy female smokers across the menstrual cycle and to compare their GABA levels with those from a healthy female non-smoking control group. | 8 weeks
  To measure occipital cortex GABA concentrations in healthy female smokers across the menstrual cycle and to compare their GABA levels with those from a healthy female non-smoking control group.
To determine the impact of 10-14 days of smoking abstinence on cortical GABA concentrations in female smokers. | 10-14 days
  To determine the impact of 10-14 days of smoking abstinence on cortical GABA concentrations in female smokers.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia N Epperson, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Center for Women's Behavioral Wellness, University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Epperson CN, Haga K, Mason GF, Sellers E, Gueorguieva R, Zhang W, Weiss E, Rothman DL, Krystal JH. Cortical gamma-aminobutyric acid levels across the menstrual cycle in healthy women and those with premenstrual dysphoric disorder: a proton magnetic resonance spectroscopy study. Arch Gen Psychiatry. 2002 Sep;59(9):851-8. doi: 10.1001/archpsyc.59.9.851. PMID 12215085
- [Background] Epperson CN, O'Malley S, Czarkowski KA, Gueorguieva R, Jatlow P, Sanacora G, Rothman DL, Krystal JH, Mason GF. Sex, GABA, and nicotine: the impact of smoking on cortical GABA levels across the menstrual cycle as measured with proton magnetic resonance spectroscopy. Biol Psychiatry. 2005 Jan 1;57(1):44-8. doi: 10.1016/j.biopsych.2004.09.021. PMID 15607299
- [Background] Epperson CN, Toll B, Wu R, Amin Z, Czarkowski KA, Jatlow P, Mazure CM, O'Malley SS. Exploring the impact of gender and reproductive status on outcomes in a randomized clinical trial of naltrexone augmentation of nicotine patch. Drug Alcohol Depend. 2010 Nov 1;112(1-2):1-8. doi: 10.1016/j.drugalcdep.2010.04.021. Epub 2010 Jun 19. PMID 20561758
- See also: Program Website — http://www.med.upenn.edu/womenswellness/